CLINICAL TRIAL: NCT00003276
Title: A Phase II Study of CPT-11 in Patients With Advanced Gallbladder or Bile Duct Tumors
Brief Title: Irinotecan in Treating Patients With Advanced Gallbladder or Bile Duct Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-964252; CDR0000066181 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Gallbladder Cancer
Keywords: unresectable gallbladder cancer; recurrent gallbladder cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan (Experimental): Patients receive a 90 minute continuous infusion of irinotecan on days 1, 8, 15, and 22 for 4 weeks, followed by a 2 week rest period. Courses of treatment are repeated every 42 days. Patients continue treatment in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year, then every 6 months for the next 4 years.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients with advanced gallbladder or bile duct cancer that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the objective tumor response rate in patients with advanced gallbladder or bile duct tumors treated with irinotecan. II. Evaluate time-to-progression, survival, and toxic effects associated with irinotecan given weekly for 4 weeks every 6 weeks in this patient population.

OUTLINE: Patients receive a 90 minute continuous infusion of irinotecan on days 1, 8, 15, and 22 for 4 weeks, followed by a 2 week rest period. Courses of treatment are repeated every 42 days. Patients continue treatment in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year, then every 6 months for the next 4 years.

PROJECTED ACCRUAL: Approximately 22-40 patients will be accrued for this study over 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven gallbladder or bile duct carcinoma with metastatic or recurrent disease deemed unresectable and not considered a candidate for potentially curative therapy Measurable or evaluable disease No known active CNS disease Closed to bile duct carcinoma as of July 1999

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT no greater than 5 times upper limit of normal (ULN) Bilirubin no greater than 1.5 mg/dL OR Bilirubin no greater than 2 times ULN in patients with biliary stents or percutaneous biliary catheters Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease Other: Nutritional intake at least 1200 kcal/day No uncontrolled infection or chronic debilitating disease Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled seizure disorder No prior malignancy within 5 years except adequately treated basal cell/squamous cell carcinomas and adequately treated noninvasive carcinomas

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biological therapy or immunotherapy for recurrent or metastatic disease No concurrent biologic therapy Chemotherapy: No prior chemotherapy for recurrent or metastatic disease Prior adjuvant chemotherapy allowed if used as a radiation sensitizer for completely resected disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for recurrent or metastatic disease Prior adjuvant radiotherapy allowed if used as a radiation sensitizer for completely resected disease No radiotherapy to greater than 25% of bone marrow No radiotherapy within the past 4 weeks No concurrent radiotherapy Concurrent CNS radiation allowed Surgery: No post abdominal exploration (with or without resection) within the past 4 weeks Other: No concurrent medication for other medical conditions except for: Analgesics Chronic treatments for preexisting conditions Agents required for life-threatening medical conditions No laxatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-03; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
objective tumor response rate | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years
time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Alberts SR, Fishkin PA, Burgart LJ, Cera PJ, Mahoney MR, Morton RF, Johnson PA, Nair S, Goldberg RM; North Central Cancer Treatment Group. CPT-11 for bile-duct and gallbladder carcinoma: a phase II North Central Cancer Treatment Group (NCCTG) study. Int J Gastrointest Cancer. 2002;32(2-3):107-14. doi: 10.1385/ijgc:32:2-3:107. PMID 12794246
- [Result] Fishkin P, Alberts S, Mahoney M, et al.: Irinotecan (CPT-11) in patients (Pts) with advanced gallbladder (GB) Carcinoma (CA): a North Central Cancer Treatment Group (NCCTG) phase II study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-618, 2001.
- [Result] Alberts S, Mahoney M, Fishkin P, et al.: Toxicity of irinotecan (CPT-11) in patients (PTS) with advanced gallbladder (GB) or biliary (BILI) tumors: a North Central Cancer Treatment Group (NCCTG) study. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-1166, 2000.